CLINICAL TRIAL: NCT07369583
Title: Monolithic Zirconia Full-Arch Rehabilitation Using a Motion-Integrated Digital Workflow Combining M-4 and All-on-4 Protocols: A Clinical Report
Brief Title: Monolithic Zirconia Full-Arch Rehabilitation Using Digital Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, Clinical Professor and principle investigator, Menoufia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADMNF-0050
Record Dates: First submitted 2025-12-02; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motion-integrated digital full-arch rehabilitation (M-4 maxilla / All-on-4 mandible) (Experimental): A fully digital, motion-integrated implant rehabilitation protocol combining the M-4 concept in the maxilla and the All-on-4 concept in the mandible. The arm included prosthetically driven planning using CBCT, intraoral and facial scanning, stackable and mucosa-supported surgical guides, immediate loading, jaw-motion tracking-guided occlusal design, and definitive monolithic zirconia full-arch prostheses connected to titanium multi-unit abutments.
  Interventions: Device: Motion-Integrated, Fully Digital Full-Arch Implant Rehabilitation Combining Maxillary M-4 and Mandibular All-on-4 Protocols with Monolithic Zirconia Prostheses

INTERVENTIONS:
Device: Motion-Integrated, Fully Digital Full-Arch Implant Rehabilitation Combining Maxillary M-4 and Mandibular All-on-4 Protocols with Monolithic Zirconia Prostheses — Participants will undergo full-arch implant rehabilitation using a fully digital, motion-integrated workflow. In the maxilla, the M-4 protocol will guide anterior implant placement in areas of limited bone, while the mandible will be rehabilitated using the All-on-4 concept with tilted posterior implants. Dual-scan CBCT and facial scans will enable prosthetically driven planning, and surgical guides-stackable in the maxilla and mucosa-supported in the mandible-will ensure precise implant placement. Real-time mandibular motion data will be incorporated into the CAD design to optimize occlusion. Definitive monolithic zirconia prostheses will be fabricated and delivered on titanium multi-unit abutments using Rosen screws, providing immediate, rigid, and esthetic full-arch restoration.

SUMMARY:
20 edentulous patients presented for full-arch rehabilitation and was managed using a motion-integrated, fully digital workflow that combined the M-4 protocol in the maxilla with the All-on-4 concept in the mandible. Dual-scan CBCT and facial scans enabled prosthetically driven planning, while stackable and mucosa-supported surgical guides facilitated precise implant placement. Real-time jaw-motion data were incorporated into the design process to individualize occlusion, and definitive monolithic zirconia prostheses were fabricated and delivered on titanium multi-unit abutments using Rosen screws.

DETAILED DESCRIPTION:
20 edentulous patients sought comprehensive full-arch rehabilitation to improve function, esthetics, and overall oral comfort. Management was performed using a fully digital, motion-integrated workflow that strategically combined two established implant protocols: the M-4 technique in the maxilla to maximize anterior anchorage in areas of limited bone volume, and the All-on-4 concept in the mandible to provide stable posterior support with tilted distal implants. Treatment planning began with dual-scan CBCT imaging and high-resolution facial scans, allowing accurate alignment of skeletal, dental, and soft-tissue datasets for prosthetically driven virtual design. A stackable guide system was employed in the maxilla to sequentially guide fixation, osteotomy preparation, and implant placement, whereas a mucosa-supported guide was used in the mandible to ensure stable positioning on the residual ridge. During the prosthetic phase, real-time mandibular motion was recorded and integrated into the CAD software to refine occlusal morphology according to the patient's functional movements. Definitive monolithic zirconia full-arch prostheses were then digitally fabricated and secured to titanium multi-unit abutments using Rosen screws, providing a rigid, precise, and metal-free restorative solution. This coordinated workflow addressed both functional and esthetic demands, enabling an efficient, patient-specific approach to immediate full-arch rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-65 years with edentulism in one or both arches.
* Adequate bone volume in the anterior maxilla for M-4 protocol and mandible for All-on-4 placement.
* Willingness to undergo full-arch implant rehabilitation using a digital workflow.
* Ability to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Systemic conditions contraindicating implant surgery (e.g., uncontrolled diabetes, immunosuppression).
* Active oral infections or untreated periodontal disease.
* Heavy smokers (>10 cigarettes/day) or substance abuse.
* History of head and neck radiation therapy or bisphosphonate use.
* Pregnancy or breastfeeding.

Ages: 40 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss | 12 months post-implant placement
  Marginal bone loss will be evaluated using periapical radiographs

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No
Up on reasonable request